CLINICAL TRIAL: NCT02651701
Title: Preoperative Imaging for Rectal Cancer Staging Using Whole Body MR-PET
Brief Title: Rectal Cancer Staging Using Whole Body MR-PET
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Jeong Hee Yoon, MD, Seoul National University Hospital
Other Study IDs: MRPET-CRC
Record Dates: First submitted 2016-01-05; First posted 2016-01-11 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: MR-PET — whole body MR-PET with dedicated liver+rectal protocol

SUMMARY:
The purpose of this study is to measure the diagnostic performance of whole body (WB) MR-PET for staging rectal cancer, compared with current standard of care (chest/abdominopelvic CT and rectal MRI) to investigate clinical feasibility of WB MR-PET as a one-stop preoperative imaging modality in patients with rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients newly diagnosed with rectal cancer on colonoscopy or sigmoidoscopy, who are potentially eligible for neoadjuvant chemoradiotherapy.
2. Patients who sign informed consent.

Exclusion Criteria:

1. Patients who are contraindication for CECT
2. Patients who are contraindication for MRI/CE-MRI
3. patients who are diagnosed with Tis or T1 cancer after polypectomy or EMR
4. Patients who were already diagnosed with an active other cancers.
5. Premenopausal female patients who are pregnant.
6. Patients with fasting serum glucose level (>200mg/dL) on blood glucose meter prior to WB MR-PET.
7. Patients who are physically compromised to undergo WB MR-PET.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients newly diagnosed with rectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-08-08 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
the concordance rate between rectal cancer staging performed by WB MR-PET and the current standard of care (chest/abdominopelvic CT and rectal MRI | 12 months
  the concordance rate between two protocols (standard protocol vs. WB-MR-PET) would be calculated.

SECONDARY OUTCOMES:
incidence of recommendation for further workup after examination | 12 months
  incidence of recommendation for further w/u after two protocols (standard vs. study) would be compared.
concordance rate of clinical staging between standard of care and that obtained by combination of WB MR-PET and chest CT. | 12 months
concordance rate of clinical stagings and true M staging obtained by biopsy or follow-up | 18 months

OTHER OUTCOMES:
Transient dyspnea | within an hour after MR contrast media administration
  incidence of transient dyspnea which can occur after MR contrast agent administration and spontaneously regressed.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong Hee Yoon, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yoon JH, Lee JM, Chang W, Kang HJ, Bandos A, Lim HJ, Kang SY, Kang KW, Ryoo SB, Jeong SY, Park KJ. Initial M Staging of Rectal Cancer: FDG PET/MRI with a Hepatocyte-specific Contrast Agent versus Contrast-enhanced CT. Radiology. 2020 Feb;294(2):310-319. doi: 10.1148/radiol.2019190794. Epub 2019 Dec 3. PMID 31793850